CLINICAL TRIAL: NCT01821846
Title: A 6-month, Multi-centre, Open Labelled, Non-randomized, Non-interventional, Safety Study of Liraglutide (Victoza®) in Subjects With Type 2 Diabetes Mellitus in Korea
Brief Title: Investigating the Safety Profile of Liraglutide Under Normal Conditions of Use in Korean Subjects With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-3929; U1111-1132-2221 (Other: WHO)
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liraglutide
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Administered either alone or in combination therapy according to the package insert (PI). Self-administered once daily, at any time subcutaneously (s.c., under the skin) in the abdomen, thigh or upper arm).

SUMMARY:
This trial is conducted in Asia. The aim of this study is to investigate the safety profile of liraglutide (Victoza®) under normal conditions of use in Korean subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with T2DM (Type 2 Diabetes Mellitus), including newly-diagnosed subjects, who require treatment with Victoza® according to the clinical judgment of their treating physician
* Subjects (and/or parents or the subject's legally acceptable representative) who are capable of giving study-specific signed informed consent before any collection of information

Exclusion Criteria:

* Subjects with a hypersensitivity to Victoza® or to any of the excipients
* Subjects who are pregnant, breast feeding or have the intention of becoming pregnant within the study periods
* Subjects with personal or family history of medullary thyroid carcinoma (MTC)
* Subjects with multiple endocrine neoplasia syndrome type 2 (MEN2)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Victoza® will be prescribed and titrated by the physician.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
The incidence of SADRs (Serious Adverse Drug Reactions) | Up to 6 months

SECONDARY OUTCOMES:
HbA1c (Glycosylated haemoglobin) change | Month 0, month 6
Percentage of subjects reaching the target of HbA1c below 7.0% | Month 6
Change in body weight | Month 0, month 6
Number of SAEs/ ADRs (Serious Adverse Events/Adverse Drug Reactions) | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- South Korea (4):
  - Novo Nordisk Investigational Site, Pyungchon-Dong 896, Dongan-Gu
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Ulsan
  - Novo Nordisk Investigational Site, Wŏnju

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com